CLINICAL TRIAL: NCT04459767
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY OPEN, PLACEBO-CONTROLLED, SINGLE ASCENDING DOSE STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF-07285557 (VUPANORSEN) ADMINISTERED SUBCUTANEOUSLY IN JAPANESE HEALTHY ADULTS WITH ELEVATED TRIGLYCERIDES
Brief Title: Investigation Of Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single Doses Of Vupanorsen In Japanese Healthy Adult Participants With Elevated Triglycerides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C4491006
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: Triglycerides
MeSH Terms: interventions — vupanorsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Vupanorsen 80 milligram (mg) (Experimental): Participants will receive one, 0.8 milliliter (mL) subcutaneous injection with vupanorsen 100 mg/mL solution
  Interventions: Drug: Vupanorsen
- Vupanorsen 160 mg (Experimental): Participants will receive two, 0.8 mL subcutaneous injections with vupanorsen 100 mg/mL solution
  Interventions: Drug: Vupanorsen
- Placebo (Placebo Comparator): Participants in Cohort 1 (vupanorsen 80 mg) will receive one 0.8 mL subcutaneous injection with 0.9% sodium chloride in water.
  Participants in Cohort 2 (vupanorsen 160 mg) will receive two 0.8 mL subcutaneous injections with 0.9% sodium chloride in water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vupanorsen — 80 mg subcutaneous injection
  Arms: Vupanorsen 160 mg; Vupanorsen 80 milligram (mg)
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double blind, third party open (i.e., participant blind, investigator blind and sponsor open), placebo controlled, single ascending dose study to investigate the safety, tolerability, pharmacokinetic and pharmacodynamics of vupanorsen in Japanese healthy adult participants with elevated triglycerides.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 20 to 65 years of age, inclusive, at the time of signing the ICD.
2. Participants must have four Japanese grandparents born in Japan.
3. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests (except for TG levels), and 12 lead ECG monitoring.
4. Fasting TG >= 90 mg/dL at Screening
5. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
6. BMI of 17.5 to 35.0 kg/m2; and a total body weight >50 kg (110 lb)
7. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
2. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb.
3. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. History of allergic or anaphylactic reaction.
5. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
6. Previous administration with an investigational drug within 4 months or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
7. A positive urine drug test.
8. Screening supine BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
9. Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
10. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level >=1.25 × ULN;
    * Total bilirubin level >=1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is=<ULN.
11. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
12. Blood donation (excluding plasma donations and platelet donations) of approximately 400 mL within 3 months or >=200 mL within a month prior to dosing. Additionally, approximately >=400 mL within 4 months for female participants.
13. History of sensitivity to heparin or heparin induced thrombocytopenia.
14. History of substance abuse within 12 months of the screening visit.
15. Pregnant females; breastfeeding females.
16. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
17. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | Day 0-90
Incidence of abnormal and clinically relevant changes in electrocardiogram | Day 0-90
Incidence and magnitude of abnormal laboratory findings | Day 0-90
Incidence of abnormal and clinically relevant changes in pulse rate | Day 0-90
Incidence of abnormal and clinically relevant changes in supine blood pressure | Day 0-90

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 0-90
Time to reach maximum observed plasma concentration (Tmax) | Day 0-90
Area under the plasma concentration-time profile from time zero to 24 hours post-dose (AUC24h) | Day 0-90
Area under the plasma concentration-time profile from time zero to 48 hours post-dose (AUC48h) | Day 0-90
Area under the plasma concentration-time profile from time zero to the last measurable concentration (AUClast) | Day 0-90
Area under the plasma concentration-time profile from time zero to infinity (AUCinf) | Day 0-90
Terminal elimination half life (t1/2) | Day 0-90
Apparent volume of distribution (Vz/F) | Day 0-90
Apparent clearance (CL/F) | Day 0-90
Percentage changes from baseline in serum angiopoietin-like protein 3 | Day 0-90
Percentage changes from baseline in total cholesterol | Day 0-90
Percentage changes from baseline in low density lipoprotein cholesterol | Day 0-90
Percentage changes from baseline in non-high-density lipoprotein cholesterol | Day 0-90
Percentage changes from baseline in very low density lipoprotein cholesterol | Day 0-90
Percentage changes from baseline in triglyceride | Day 0-90
Percentage changes from baseline in apolipoprotein A-1 | Day 0-90
Percentage changes from baseline in apolipoprotein B total | Day 0-90
Percentage changes from baseline in apolipoprotein C-III | Day 0-90

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one Clinic, Hachioji-shi, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Fukuhara K, Furihata K, Matsuoka N, Itamura R, Ramos V, Hagi T, Kalluru H, Bramson C, Terra SG, Liu J. A multi-purpose Japanese phase I study in the global development of vupanorsen: Randomized, placebo-controlled, single-ascending dose study in adults. Clin Transl Sci. 2023 May;16(5):886-897. doi: 10.1111/cts.13498. Epub 2023 Mar 31. PMID 37002654
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4491006